CLINICAL TRIAL: NCT04821440
Title: A 3D Tablet Sensor Approach to the Measurement of an Upper and Lower Limb Volume in the Monitoring of a Lymphedema
Brief Title: A 3D Tablet Sensor Approach to the Measurement of a Lymphedema
Acronym: LO3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 29BRC20.0049
Record Dates: First submitted 2020-05-26; First posted 2021-03-29 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Lymphedema
Keywords: 3D sensor; Lower Extremity; Upper Extremity; Body Regions; Measurement; Monitoring; Water displacement; Volume
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower Limb Lymphedema (Active Comparator): Patients suffering from unilateral lower-limb lymphedema will receive volume measurements of their limb three times, once with the water displacement method, twice with the 3D sensor method
  Interventions: Device: Water displacement volumetry; Device: Three dimension volumetry
- Upper Limb Lymphedema (Active Comparator): Patients suffering from unilateral upper-limb lymphedema will receive volume measurements of their limb three times, once with the water displacement method, twice with the 3D sensor method
  Interventions: Device: Water displacement volumetry; Device: Three dimension volumetry

INTERVENTIONS:
Device: Water displacement volumetry — The examination will take place in several stages and by two operators. Initially, the patient will strip the limb concerned (leg or arm). Once the member is in the water column of the volumeter, a delimitation of the submerged area of the member will be carried out using a marking (black dermographic marker). Indeed, the level of acquisition in 3D is determined relative to the height of the water line marked on the skin with a black felt, this felt is usually used for venous mapping and is well tolerated The first operator will carry out two measurements one after the other with a change of water previously stabilized at room temperature.
Device: Three dimension volumetry — The 3D volumetric acquisition is done with the sensor (CE marking) attached to the touch pad and does not require invasive or cutaneous contact with the patient (minimum acquisition distance of 40 cm). The operator triggers the acquisition via a button in an application installed on the tablet and physically turns around the patient to carry out the acquisition of the affected member. At the end of the acquisition, the operator presses a stop button and chooses whether or not to calculate the volume using another button depending on the quality of the acquisition.

SUMMARY:
Up to now, the diagnosis of lymphedema remains hard and delayed. It suffers from many limitations such as lack of coordination and formation of the health-care network. The diversity of used tools is another obstacle because all provided solutions on the market are either costless with poor accuracy, or highly expensive but with excellent accuracy. Therefore, we decided to evaluate an affordable and open-source 3D iPad sensor sharing the same technology used in Kinect sensors.

ELIGIBILITY:
Inclusion Criteria:

- Unilateral lymphedema

Exclusion Criteria:

* Minor patient,
* Bilateral lymphedema,
* Trophic disorders: Acute or recent skin infection (<1 month after the end of antibiotic therapy), unhealed wounds.
* Predictable difficulties in carrying out the measurements due to the patient's physical limitations (maintenance of orthostatic or sitting position <5 minutes)
* Single or bilateral edema with a different etiology than lymphedema.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Accuracy of a 3D sensor for lymphedema volumetry | One hour
  Intra-class correlation coefficient (ICC) Mean bias and limits of agreement (LOA) derived from the Blant-Altman diagram Mean bias and limits of agreement (LOA) derived from the Blant-Altman diagram

SECONDARY OUTCOMES:
Reproducibility of measurements made with a 3D sensor for lymphedema volumetry | One hour
  Intra-class correlation coefficient (ICC)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Brest, Brest
  - CH Pont l'Abbé, Pont-l'Abbé